CLINICAL TRIAL: NCT00115804
Title: An Open-Label Clinical Trial of Fluoxetine Treatment of Juvenile Primary Fibromyalgia Syndrome
Brief Title: Safety and Efficacy of Fluoxetine in Juvenile Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Lesley M. Arnold, M.D., Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-3-22-1
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Juvenile Primary Fibromyalgia Syndrome (JPFS); Fibromyalgia
Keywords: Fibromyalgia; Juvenile
MeSH Terms: conditions — Fibromyalgia | interventions — Fluoxetine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine (Experimental): All eligible patients were started on Fluoxetine at 10 mg once daily. The dose was flexibly dosed based on pain efficacy and tolerability to a final dose between 10 and 60 mg once daily.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine po 10-60 mg/day for 12 weeks. Fluoxetine was started at 10 mg once daily. The dose was flexibly dosed based on pain efficacy and tolerability to a final dose between 10 and 60 mg once daily
  Other Names: Prozac

SUMMARY:
The purpose of this research is to conduct an open, pilot trial to assess the efficacy and safety of fluoxetine in the treatment of Juvenile Primary Fibromyalgia Syndrome (JPFS).

DETAILED DESCRIPTION:
Fibromyalgia is a common condition that is often challenging to treat. It is defined by the American College of Rheumatology (ACR) as widespread pain of at least 3 months duration in combination with tenderness at 11 or more of 18 specific tender point sites on the body. The prevalence of JPFS in children and adolescents in the general population of the United States is unknown. Studies from Israel, Mexico, and Italy have estimated that the prevalence rate of JPFS in school children ranges from 1.24% to 6.20%, with girls making up the majority of cases. Information from a national registry in the United States indicates that JPFS accounts for about 7.7% of new patient diagnoses in a pediatric rheumatology setting. The mean age of onset of pediatric JPFS is 12 years. As in adults, JPFS has been diagnosed in children and adolescents using the ACR criteria. JPFS often leads to substantial morbidity and disability. For example, adolescents with JPFS reported significantly greater functional disability and greater number of school absences than those with other rheumatic diseases such as juvenile RA or lupus. The presence of high levels of pain and disability at this critical developmental stage place adolescents with JPFS at greater risk for long term social and occupational difficulties. Early diagnosis and effective intervention are therefore of critical importance.

ELIGIBILITY:
Inclusion Criteria:

* Female or male outpatients 13 to 18 years of age.
* Fulfillment of the American College of Rheumatology (ACR) criteria for primary fibromyalgia.
* Ability to understand and cooperate with study procedures.
* Provision of parental written informed consent and verbal and written assent from the adolescent for participation in the study.

Exclusion Criteria:

* Unwillingness or inability on the part of the parent to provide written informed consent or for the adolescent to provide verbal and written assent.
* Lifetime history of psychosis, hypomania or mania.
* Diagnosis of alcohol or substance abuse or dependence within 6 months prior to screening visit.
* Patients judged to be at serious suicide or homicide risk.
* Girls who are pregnant or lactating. Girls of childbearing potential who are not using a medically accepted method of contraception (including barrier or hormonal methods).
* Clinically unstable medical or psychiatric conditions that could interfere with the absorption, metabolism, excretion, or safety of fluoxetine or interfere with the assessment of disease severity.
* Inability to exclude traumatic injury, regional or structural rheumatic disease, or infectious arthropathy as the etiology of their relevant fibromyalgia symptoms and that would interfere with interpretation of outcome measures (e.g., osteoarthritis, bursitis, tendonitis).
* History of an autoimmune disease or inflammatory arthritis, such as systemic lupus erythematosis (SLE) or rheumatoid arthritis (RA).
* Treatment with a monoamine oxidase inhibitor, tricyclic, selective serotonin reuptake inhibitor (SSRI) antidepressant, or lithium within 2 weeks prior to beginning study medication.
* Treatment with analgesic medication (with the exception of acetaminophen and over-the-counter NSAIDs) within one week prior to beginning study medication.
* Treatment with any other excluded medication that cannot be discontinued at the screening visit.
* Previous treatment with fluoxetine.
* Treatment with any investigational medications within 30 days prior to screening.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2005-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley M Arnold, M.D., Principal Investigator — Women's Health Research Program
Locations (1):
- Women's Health Research Program, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female or male patients from Children's Hospital pediatric outpatient rheumatology clinic were eligible for the trial if they were 13 to 17 years and met study criteria.
Pre-assignment Details: Patients who met entry criteria for juvenile fibromyalgia but did not meet any exclusion criteria.
Groups:
- Fluoxetine: All patients receiving Fluoxetine starting at 10 mg/day
Period: Overall Study
Arm/Group | Fluoxetine
Started | 6
Completed | 4
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Fluoxetine: All eligible patients were given fluoxetine
Arm/Group | Fluoxetine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Average Pain Severity [Mean (Full Range); unit: mm] — The average pain severity on the Pediatric Pain Questionnaire's 100-mm visual analog scale. This is a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of zero "no pain at all" and 100 "worst pain imaginable."
  mm | 62 [47 to 76]

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Severity Score
Description: The primary outcome measure was average pain severity on the Pediatric Pain Questionnaire's 100-mm visual analog scale.
  (0=no pain and 100 = severe pain )
Time Frame: Daily on average in the past week.
Population: 6 participants out of 10 screened met entry criteria. Two were terminated due to serious adverse events (SAEs).
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Fluoxetine: Fluoxetine was started at 10 mg/day and adjusted based on pain efficacy and tolerability.
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
mm | 62 (11.9)

2. Secondary Outcome: The Clinical Global Impression of Severity
Description: Measures severity of illness at the time of the assessment on a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill).
Time Frame: at the time of the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluoxetine: All eligible patients were started on Fluoxetine at 10 mg once daily. The dose was flexibly dosed based on pain efficacy and tolerability to a final dose between 10 and 60 mg once daily.
  Fluoxetine: fluoxetine po 10-60 mg/day for 12 weeks
  Fluoxetine: Fluoxetine was started at 10 mg once daily. The dose was flexibly dosed based on pain efficacy and tolerability to a final dose between 10 and 60 mg once daily.
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 5 (1.1)

3. Secondary Outcome: The Patient Global Impression of Improvement
Description: Measures the patient's impression of improvement since baseline on a scale of 1 (very much better) to 7 (very much worse).
Time Frame: since baseline, at the time of the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 1.5 (0.5)

4. Secondary Outcome: The Functional Disability Inventory-child Version
Description: A self-report inventory that assesses patients' ability to perform a variety of daily physical, social, and recreational activities. The scale ranges from 0 (no disability) to 60 (severe disability).
Time Frame: Over the "last few days."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 24.2 (12.5)

5. Secondary Outcome: The Functional Disability Inventory-parent Version
Description: Consists of the same 15 items as the child version but allows the parent to provide their perception of the child's difficulty in performing daily physical, social, and recreational activities. The score ranges from 0 (no disability) to 60 (severe disability).
Time Frame: Over the "last few days."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 19.2 (12.4)

6. Secondary Outcome: Children's Depression Inventory
Description: A 27-item, self-report measure of depressive symptoms with a score range of 0 (no depressive symptoms) to 54 (severe depressive symptoms.
Time Frame: Over the past 2 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 14.2 (10.3)

7. Secondary Outcome: Multidimensional Anxiety Scale for Children
Description: A 39-item self-report inventory that assesses four areas of anxiety symptoms (emotional, cognitive, physical, and behavioral). Score ranges from 0 (no anxiety symptoms) to 117 (severe anxiety symptoms).
Time Frame: Over the past week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 52 (30.9)

8. Secondary Outcome: Fibromyalgia Impact Questionnaire Modified for Children
Description: A 19 item self-report instrument that measures overall impact of fibromyalgia including assessments of function, pain, fatigue, sleep quality, stiffness, anxiety and depression. Score range from 0 (no impact) to 100 (severe impact).
Time Frame: Over the past week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 4
units on a scale | 55.1 (23.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Period after screening when fluoxetine was started
Arm/Group | Fluoxetine
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=6)
Viral Adenitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=6)
Headache (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes